CLINICAL TRIAL: NCT04550260
Title: A Phase III, Randomized, Double-Blind, Placebo Controlled, Multi-Center, International Study of Durvalumab Given Concurrently With Definitive Chemoradiation Therapy in Patients With Locally Advanced, Unresectable Esophageal Squamous Cell Carcinoma (KUNLUN)
Brief Title: Study of Durvalumab Versus Placebo in Combination With Definitive Chemoradiation Therapy in Patient With ESCC
Acronym: KUNLUN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D910SC00001; 2020-001001-22 (EudraCT Number)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Locally Advanced unresectable ESCC; PD-L1; Durvalumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — durvalumab; CF regimen; Cisplatin; Capecitabine; Radiation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor, excluding supply chain management personnel, will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Durvalumab + definitive CRT (Experimental): Durvalumab + concurrent chemoradiation
  Interventions: Drug: Durvalumab; Drug: cisplatin + fluorouracil; Drug: cisplatin + capecitabine; Radiation: Radiation
- Arm 2: Placebo + definitive CRT (Placebo Comparator): Placebo + concurrent chemoradiation
  Interventions: Drug: Placebo; Drug: cisplatin + fluorouracil; Drug: cisplatin + capecitabine; Radiation: Radiation

INTERVENTIONS:
Drug: Durvalumab — Durvalumab intravenous infusion
  Other Names: MEDI4736
  Arms: Arm 1: Durvalumab + definitive CRT
Drug: Placebo — Durvalumab matching placebo for intravenous infusion
  Arms: Arm 2: Placebo + definitive CRT
Drug: cisplatin + fluorouracil — cisplatin + fluorouracil, as per Standard of Care
Drug: cisplatin + capecitabine — cisplatin + capecitabine, as per Standard of Care
Radiation: Radiation — 50-64Gy in total

SUMMARY:
This is a Phase III, randomized, double-blind, placebo-controlled, multi-center international study to assess the efficacy and safety of durvalumab administered concurrently with dCRT in patients with locally advanced, unresectable esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
Approximately 600 patients with locally advanced, unresectable ESCC (AJCC 8th cStage II-IVA) will be randomized in a 2:1 ratio to receive either durvalumab + dCRT or placebo + dCRT. The primary objectives of this study are to assess the efficacy of durvalumab + dCRT compared with placebo + dCRT in terms of progression free survival (PFS, per RECIST 1.1 as assessed by BICR) in PD-L1 High population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of signing the ICF.
* Histologically or cytologically confirmed esophageal squamous cell carcinoma, and present with locally advanced disease (Stage II-IVA).
* Unresectable or refusing surgery, and has been deemed suitable for definitive chemoradiation therapy.
* Patients with at least an evaluable lesion per RECIST 1.1.
* Mandatory provision of available tumor tissue for PD-L1 expression analysis.
* ECOG PS 0 or 1.
* Adequate organ and marrow function.
* Life expectancy of more than 3 months.

Exclusion Criteria:

* Histologically or cytologically confirmed small cell esophageal carcinoma, esophageal adenocarcinoma or other mixed carcinoma.
* Prior anti-cancer treatment for ESCC.
* Patient with a great risk of perforation and massive bleeding.
* History of allogeneic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders.
* Uncontrolled intercurrent illness.
* History of another primary malignancy.
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) per RECIST 1.1 as assessed by BICR | up to approximately 56 months
  To assess the efficacy in terms of PFS in PD-L1 High population

SECONDARY OUTCOMES:
Overall survival (OS) | up to approximately 72 months
  To assess the efficacy in terms of OS in all randomized patients and in PD-L1 High population until the date of death
Progression free survival (PFS) per RECIST 1.1 as assessed by BICR | up to approximately 56 months
  To assess the efficacy in terms of PFS in all randomized patients.

OTHER OUTCOMES:
Adverse events (AEs) | up to approximately 72 months
  To assess the safety and tolerability profile of durvalumab + dCRT compared to placebo + dCRT in patients with ESCC

CONTACTS AND LOCATIONS:
Overall Officials: Luhua Wang, MD, Principal Investigator — Cancer Hospital of Chinese Academy of Medical Science; Nabil Saba, MD, Principal Investigator — Department of Hematology and Medical Oncology, Emory University
Locations (115):
- United States (5):
  - Research Site, Atlanta, Georgia
  - Research Site, Louisville, Kentucky
  - Research Site, Dallas, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Morgantown, West Virginia
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Liège
  - Research Site, Namur
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, Vitória
- Canada (2):
  - Research Site, Barrie, Ontario
  - Research Site, Greater Sudbury, Ontario
- China (26):
  - Research Site, Anyang
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changsha
  - Research Site, Changzhi
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Huai'an
  - Research Site, Jieyang
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Liangyugang
  - Research Site, Nantong
  - Research Site, Qingdao
  - Research Site, Quanzhou
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
  - Research Site, Zhenjiang
- France (8):
  - Research Site, Besançon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Villejuif
- Japan (18):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Maebashi
  - Research Site, Matsuyama
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Yokohama
- Mexico (5):
  - Research Site, Chihuahua City
  - Research Site, Cuernavaca
  - Research Site, Mérida
  - Research Site, Monterrey
  - Research Site, Veracruz
- Poland (5):
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Siedlce
  - Research Site, Warsaw
- Russia (8):
  - Research Site, Chelyabinsk
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
  - Research Site, Tyumen
  - Research Site, Ufa
  - Research Site, Yekaterinburg
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Santander
  - Research Site, Zaragoza
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chanthaburi
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Turkey (Türkiye) (6):
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Erzurum
  - Research Site, Goztepe Istanbul
  - Research Site, Izmir
  - Research Site, Van
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home